CLINICAL TRIAL: NCT03490773
Title: Assessing Genetic and Immunological Predictors of Endogenous Insulin Production in Type 1 Diabetes
Brief Title: Type 1 Diabetes, Immunology, Genetics & Endogenous Insulin Production
Acronym: TIGI
Status: Completed | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: Leiden University Medical Center (Other); King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: CRF142; 141756 (Other: IRAS); 13/SW/0312 (Other: Research Ethics Committee)
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Cpeptide; Immunology
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cells (PBMCs) DNA Serum Plasma Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Type I diabetes(T1D)T occurs when an individual loses the ability to make enough insulin to control their blood sugar levels. They need insulin injections to replace the insulin production that has been lost. Traditionally people with T1D are thought to make none of their own insulin after diagnosis, but we have recently identified that there are some people who have T1D but go one making insulin for many years. We would like to explore this in more depth and understand why some people with T1D go on making insulin and some do not. This will help us understand the causes of T1D and may help work out ways to protect this remaining insulin production, with improved blood sugar control, and reduced long-term complications of diabetes We aim to explore genetic and immunological factors which impact on the ability of an individual diagnosed with Type I diabetes (T1D) to produce their own insulin. We aim to study individuals who have been diagnosed with T1D with variable duration and assess the genetic and immunological profile of those whose are thought to be producing significant amounts of insulin despite a long duration and those who despite a very short duration, lose insulin production very quickly.

DETAILED DESCRIPTION:
Background & Introduction:

Type 1 Diabetes (T1D) is a disease caused by the autoimmune destruction of pancreatic beta cells. It commonly presents in childhood with elevated blood sugars and long-term insulin treatment is required. People diagnosed with T1D have some pancreatic beta cells remaining at diagnosis and these remaining insulin producing cells were thought to be lost within the first few months or years after diagnosis. The underlying mechanism for destruction of beta cells is T-cell driven autoimmunity with genetic, environmental and immune associations that point towards the immune system as being the key to pancreatic beta cells loss. Extensive research has focussed on trying to prevent, halt or reverse immune attack in T1D using immunosuppression or immunomodulation with a variety of drugs and vaccines. These efforts have been largely unsuccessful and demonstrate that although we know that autoimmunity is critical to the development of T1D we still do not know enough about specific mechanisms to successfully stop this process. By better understanding the role of the immune system in T1D, this may ultimately lead to better treatments or reversal of T1D.

Contrary to conventional understanding, not all people with T1D lose insulin production soon after diagnosis. Modern assays that can detect low levels of endogenous insulin have shown that many people with T1D make low levels of insulin for many years after diagnosis. There are also a smaller group of patients who make significant amounts of insulin despite having T1D for many years. Conversely, there are some patients who seem to lose all endogenous insulin very quickly after diagnosis.

Urine C-peptide Creatinine ratio is a new technique that allows assessment of endogenous insulin production in a urine sample that is posted from home. This has allowed the assessment of insulin production in over 1000 patients with T1D in the South West of England with identification of patients still making significant amounts of insulin after years of T1D, and other patients who have lost insulin production very rapidly.

Retained endogenous insulin production may represent a slower autoimmune process, with a dampening of the immune response by regulation within the autoimmune system (tolerance), or a "burning out" of the process of autoimmunity as can happen in some other autoimmune diseases. Similarly, very rapid loss of insulin production may represent the opposite, more aggressive end of the spectrum.

We aim to study this by comparing immunological characteristics of patients with T1D, with a range of diabetes duration, and still making significant insulin with similar groups who are making none.

Hypotheses:

People with long duration T1D and maintained endogenous insulin production have an altered balance of islet destructive T cells (islet-specific auto reactive CD4 helper and CD8 killer T cells) and islet protective T cells (regulatory T-cells) and may have different genetic risk factors for autoimmune disease.

Study Aim:

To improve our understanding of insulin production in individuals diagnosed with Type 1 diabetes.

TIGI is an observational case control study. All potential participants will be identified from either routine clinical care or from existing research cohorts managed by the Peninsula Research Bank as part of the NIHR Exeter Clinical Research Facility (ECRF). Potential participants who appear to meet the entry criteria will be given written information on the project, followed by the opportunity to discuss the project in more detail with a member of the research team. The research team will be responsible for the recruitment process.

Participants will be recruited under UK wide ethics.

All participants (or their legal guardians) will be required to provide written informed consent and will be informed of their right to withdraw from the stud at any time with prejudice or jeopardy to any future clinical care.

Participants will be asked to attend the NIHR Exeter Clinical Research Facility for a single appointment, having fasted overnight. To reduce patient burden, participants who are unable to visit the research facility will be offered an appointment locally (e.g. home or GP surgery). They will have been asked to provide a urine sample to be collected 2 hours after their main meal on the day before the study visit (for analysis of UCPCR).

Blood samples will be collected at baseline (fasting) and at 0, 30,60, 90 & 120 minutes post meal for adult participants attending the research facility. For children under 16 years of age and all participants recruited at home, samples will be collected at 90 minutes post meal only.

Baseline data will include: Height (m), weight (kg), age of diagnosis, current and previous insulin treatment and family history of diabetes.

Blood samples will be collected for Serum C-peptide and other routine biochemistry, DNA extraction (for HLA typing and T1D risk SNP typing), Peripheral blood mononuclear cells (PBMCs) for analysis of auto reactive and regulatory T-cells, and plasma and serum samples for storage for future analysis.

All samples will be appropriately labelled in accordance with the 1998 Data Protection Act. Biological samples collected from participants will be transported, stored, accessed and processed in accordance with national legislation relating to the use and storage of human tissue for research purposes. Participants will have the opportunity to consent to gift samples at the end of the study for future research.

Safety: Blood samples will be collected by staff trained in venepuncture. Any potential discomfort or side -effects will be equivalent to that experienced in routine clinical care. Risk of hyperglycemia (from having a meal without their usual mealtime insulin): Participants will be closely monitored during and after their visit by the diabetes specialist research team. Appropriate advice/support will be given if required.

Potential Benefit: In the short term we hope to gain an improved understanding of the causes of T1D. In the longer term this work may lead to improved therapeutic, vaccine and transplantation treatments for T1D.

Adverse Effects: Should any unforeseen adverse events arise that possibly, probably or definitely related to a study procedure, they wil be reported to the Sponsor and CI within 24 hours of the research team becoming aware of the event.

Confidentiality: All information related to study participants will be kept confidential and managed in accordance with the Data Protection Act, NHS Caldicott Guardian, The Research Governance Framework for Health & Social Care and Research Ethics Committee Approval.

Participant date will be held in link-anonymised format, with personal identifiable data only accessible to personnel with training in data protection who require this information to perform their study role.

Record Retention & Archiving: When the research study is complete, it is a requirement of the Research Governance Framework and Sponsor Trust Policy that the records are kept for a further 15 years.

Statistics & Sample Size:

The main analysis will be to assess if there is a difference in the immune phenotype of patients with the most (High C-peptide) and the least (Low C-peptide) persistent endogenous insulin relative to duration.

We will recruit at least 110 patients in each group in keeping with previous recruitment in Exeter. We predict a minimum of 100 will have confirmed extreme C-peptide in each group. This will give 90% power to detect at p<0.01, a difference of 0.6 standard deviation in measures of immune function and a difference in proportions of 30 (50 v 80)%. Previous studies have shown differences of >1 SD in the mean suppressive function of autoreactive T cells and a difference in proportion of 39%.

The total sample size for this project will be at least 250, to achieve the required number of patients with extreme C-peptide as detailed above.

Both groups will have a range of diabetes duration.

Monitoring of this study will ensure compliance with Good Clinical Practice. The Investigators will permit monitoring, audits, REC review and regulatory inspections by providing the Sponsor(s), Regulators and REC direct access to source data and other documents.

NHS indemnity will apply to participants and UK public liability insurance is provided by the University of Exeter.

Project development and user involvement:

The study team will have access to the user representative group of the NIHR Exeter Clinical Research Facility (ECRF). In keeping with the NHS Patient Carer and Public Involvement (PCPI) strategy the ECRF invites user representatives to contribute to the development of various projects within its portfolio. These individuals have agreed to maintain contact and regular meetings have been established at which researchers discuss the development of current projects within the ECRF.

This work is funded by a patient-focused diabetes charity, JDRF. On completion of the study, the data will be analysed and a final study report will be prepared and submitted to the funder, sponsor and ethics committee. Results will be written up and submitted for publication in peer reviewed journal(s). Abstracts will be submitted to national and international conferences. Written information in the form of a letter/newsletter outlining the key findings of the study will be posted on the study web page.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 1 diabetes
* Insulin treated
* Known UCPCR status (positive/negative defined by UCPCR cut off of 0.2nmol/mmol)
* Age 5-65 years inclusive
* Able and willing to provide informed consent/assent

Exclusion Criteria:

* Pregnant or lactating (as this may limit blood sampling and affect T cell function)
* Any infectious illness within the last 2 weeks if it was a febrile illness, or within 2-3 days if it was non-febrile (as this may activate T cells non-specifically)
* Taking steroids or other immunosuppressive medications (as these may alter T cell function)
* Received any immunoglobulin treatments or blood products in the last 3 months (as these may alter T cell function)
* Any other medical condition which, in the opinion of the investigator, would affect the safety of the subject's participation.
* Recreational drug or alcohol abuse (excluding cannabis use more than 1 week prior to blood sampling) - drug abuse may alter T cell function.
* Severe complications of diabetes other than background retinopathy, uncomplicated neuropathy or proteinuria with creatinine in normal reference range (as more severe complications may affect T cell function)

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All potential participants will be identified from either routine clinical care or from existing research cohorts managed by the Peninsula Research Bank as part of the NIHR Exeter Clinical Research Facility (ECRF). Potential participants who appear to meet the entry criteria will be given written information on the project, followed by the opportunity to discuss the project in more detail with a member of the research team. The research team will be responsible for the recruitment process.
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Difference in immune function in Cpeptide negative and positive | Within 6 months of last participant visit
  The frequency or suppressive function of regulatory T-cells and the frequency of auto reactive CD4 and CD8 T cells between C-peptide positive and C-peptide negative groups, (with patients and controls individually matched for age of diagnosis and duration).

SECONDARY OUTCOMES:
Difference in HLA type in Cpeptide negative and positive groups | Within 6 months of last participant visit
  The frequency of high and low risk HLA types and the frequency of non-HLA gene polymorphisms associated with T1D risk, between C-peptide positive, and C-peptide negative groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hattersley, Professor, Principal Investigator — University of Exeter
Locations (3):
- Leiden University Medical Center, Leiden, Netherlands
- United Kingdom (2):
  - Royal Devon & Exeter NHS Foundation Trust, Exeter, Devon
  - King's College London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawson JM, Tremble J, Dayan C, Beyan H, Leslie RD, Peakman M, Tree TI. Increased resistance to CD4+CD25hi regulatory T cell-mediated suppression in patients with type 1 diabetes. Clin Exp Immunol. 2008 Dec;154(3):353-9. doi: 10.1111/j.1365-2249.2008.03810.x. PMID 19037920
- [Background] Lindley S, Dayan CM, Bishop A, Roep BO, Peakman M, Tree TI. Defective suppressor function in CD4(+)CD25(+) T-cells from patients with type 1 diabetes. Diabetes. 2005 Jan;54(1):92-9. doi: 10.2337/diabetes.54.1.92. PMID 15616015
- [Background] Hilbrands R, Huurman VA, Gillard P, Velthuis JH, De Waele M, Mathieu C, Kaufman L, Pipeleers-Marichal M, Ling Z, Movahedi B, Jacobs-Tulleneers-Thevissen D, Monbaliu D, Ysebaert D, Gorus FK, Roep BO, Pipeleers DG, Keymeulen B. Differences in baseline lymphocyte counts and autoreactivity are associated with differences in outcome of islet cell transplantation in type 1 diabetic patients. Diabetes. 2009 Oct;58(10):2267-76. doi: 10.2337/db09-0160. Epub 2009 Jul 14. PMID 19602536
- [Background] Velthuis JH, Unger WW, Abreu JR, Duinkerken G, Franken K, Peakman M, Bakker AH, Reker-Hadrup S, Keymeulen B, Drijfhout JW, Schumacher TN, Roep BO. Simultaneous detection of circulating autoreactive CD8+ T-cells specific for different islet cell-associated epitopes using combinatorial MHC multimers. Diabetes. 2010 Jul;59(7):1721-30. doi: 10.2337/db09-1486. Epub 2010 Mar 31. PMID 20357361
- [Result] Marren SM, Hammersley S, McDonald TJ, Shields BM, Knight BA, Hill A, Bolt R, Tree TI, Roep BO, Hattersley AT, Jones AG, Oram RA; TIGI consortium. Persistent C-peptide is associated with reduced hypoglycaemia but not HbA1c in adults with longstanding Type 1 diabetes: evidence for lack of intensive treatment in UK clinical practice? Diabet Med. 2019 Sep;36(9):1092-1099. doi: 10.1111/dme.13960. Epub 2019 Jun 27. PMID 30955221
- [Result] Shields BM, McDonald TJ, Oram R, Hill A, Hudson M, Leete P, Pearson ER, Richardson SJ, Morgan NG, Hattersley AT; TIGI Consortium. C-Peptide Decline in Type 1 Diabetes Has Two Phases: An Initial Exponential Fall and a Subsequent Stable Phase. Diabetes Care. 2018 Jul;41(7):1486-1492. doi: 10.2337/dc18-0465. Epub 2018 Jun 7. PMID 29880650